CLINICAL TRIAL: NCT00989339
Title: Effects of Intralipid and Olive Oil Infusion on Endothelial Function, Inflammatory Markers, Oxidative Stress, Immune Function, Autonomic Nervous System, Insulin Sensitivity and Carbohydrate Metabolism
Brief Title: Effects of Intralipid Versus Olive Oil Infusions on Endothelial Function, Immune Function, Inflammatory Markers
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sub-investigator left facility prior to study initiation
Sponsor: Emory University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00019153; IRB00019153
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes; Hypertension; Obesity
Keywords: lipid emulsion; endothelial function; inflammatory markers; oxidative stress; insulin sensitivity; carbohydrate metabolism
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Twenty-four Hour TPN and Saline Infusion (Experimental): Subjects will be admitted to the Grady research center on the evening before each study. The next morning, after an overnight fast, they will receive, in random order, Intralipid 20%, ClinOleic 20% or normal saline at 20 ml/hr for 24 hr. The interval between admissions will be 1 month.
  Interventions: Drug: Twenty-four Hour TPN and Saline Infusion

INTERVENTIONS:
Drug: Twenty-four Hour TPN and Saline Infusion — Infusion of Intralipid 20%, ClinOleic 20% or normal saline at 20 ml/hr for 24 hr.

SUMMARY:
Recent evidence suggests that increased levels of a circulation fat (free fatty acids or FFAs) can cause high blood pressure and cardiac complications. Intralipid is the only type of fat approved by the FDA for clinical use. It is usually used as nutrition support in malnourished patients. The investigators' preliminary studies indicate that Intralipid results in a significant rise in blood pressure, blood vessel stiffness, and inflammation in obese subjects. Olive oil can also be used as nutrition support. The effect of olive oil intravenous (IV) on blood pressure and inflammation is not known. In this study, the investigators will compare the effect of Intralipid and olive oil on blood pressure, blood vessel stiffness and inflammation in healthy subjects. The investigators hypothesize that Olive oil emulsions will result in less vascular changes and less inflammatory response than Intralipid solutions. Accordingly, the investigators propose a systematic evaluation of the effects of Intralipid, olive oil and normal saline on blood pressure, endothelial function (vascular stiffness), inflammation in normal subjects.

A group of obese subjects will be admitted to the Clinical Research Center on 3 occasions. Subjects will receive repeated infusions of Intralipid, ClinOleic, and normal saline at 20 ml/hour for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females
* BMI 25 -35 kg/m2, between the ages of 18 and 65 years
* BP < 140/80 mm Hg and no prior history of hypertension

Exclusion Criteria:

* Pregnancy or breast feeding
* History of diabetes, hypertension, fasting triglyceride levels > 250 mg/dL, liver disease (ALT 2.5x > upper limit of normal), serum creatinine ≥ 1.5 mg/dL, -Smokers or ex-smoker < 3 months of cessation, drug or alcohol abuse
* Mental condition rendering the subject unable to understand the scope and possible consequences of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
endothelial function | 1 year

SECONDARY OUTCOMES:
oxidative stress | 1 year
autonomic nervous system | 1 year
insulin sensitivity | 1 year
carbohydrate metabolism | 1 year